CLINICAL TRIAL: NCT06529757
Title: Skin Wetting in Burn Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STU_2020_0334_B
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Burn Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot and Dry Environment_no cooling (Experimental): Subjects will exercise for 60 minutes in a hot and dry environment while being exposed to no cooling.
  Interventions: Other: Non-cooling
- Hot and Dry Environment_whole body skin wetting (Experimental): Subjects will exercise for 60 minutes in a hot and dry environment while being exposed to whole body skin wetting.
  Interventions: Other: Whole body cooling

INTERVENTIONS:
Other: Whole body cooling — Subjects will exercise for 60 minutes in the indicated environmental condition while being exposed to whole body skin wetting. Skin wetting will be performed by spraying water onto the whole body throughout the exercise bout.
  Arms: Hot and Dry Environment_whole body skin wetting
Other: Non-cooling — Subjects will exercise for 60 minutes in the indicated environmental condition while being exposed to no cooling modalities.
  Arms: Hot and Dry Environment_no cooling

SUMMARY:
This project will identify the efficacy of whole body skin wetting aimed to attenuate excessive elevations in internal body temperatures during physical activity in well-healed burn survivors. The investigators will conduct a randomized crossover design study. Non-burned control subjects, subjects who experienced burns covering ~20% to 40% of their body surface area, and subject having burns >40% of their body surface area will be investigated. Subjects will exercise in heated environmental conditions while receiving no cooling or whole body skin wetting.

ELIGIBILITY:
Inclusion Criteria: Non-burn survivors

* Healthy male and female subjects
* 18-65 years of age.
* Free of any underlying medical conditions

Exclusion Criteria (non-burned individuals):

* Any burn-related injuries resulting in at least one night of hospitalization.
* Heart disease or any other chronic medical condition requiring regular medical therapy including cancer, diabetes, and hypertension.
* Abnormalities detected on routine screening
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2.
* Pregnant individuals

Inclusion Criteria (burn survivors):

* Healthy male and female subjects
* 18-65 years of age.
* Free of any underlying medical conditions
* Having a burn injury covering 20-40% or >40% of the participant's body surface area; at least 50% of those burn injuries must be full thickness that required skin grafting.
* Participants must have been hospitalized due to the burn injury for a minimum of 15 days

Exclusion Criteria (burn survivors):

* Any burn-related injuries resulting in at least one night of hospitalization.
* Heart disease or any other chronic medical condition requiring regular medical therapy including cancer, diabetes, and hypertension.
* Abnormalities detected on routine screening
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2.
* Pregnant individuals
* Extensive unhealed injured skin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Core Temperature | Prior to and throughout the bout of exercise; an average of 90 minutes.
  During exercise, one's core body temperature will increase. This device will measure this increase in core body temperature throughout the exercise.

SECONDARY OUTCOMES:
Mean Skin Temperature | Prior to and throughout the bout of exercise; an average of 90 minutes.
  Average skin temperature from six sites.
Rate Pressure Product | Prior to and throughout the bout of exercise; an average of 90 minutes.
  Obtained from heart rate and systolic blood pressure.
Whole body sweat rate | Before and after exercise. 2 min per measure.
  Whole body sweat rate will be measured from pre and post nude body mass measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Exercise and Environmental Medicine, Dallas, Texas, United States